CLINICAL TRIAL: NCT07034183
Title: A First-in-Human Study of PRD001 in Healthy Participants, Assessment of Safety, Tolerability and Pharmacokinetics of Single/Multiple Doses
Brief Title: A First-in-Human Study of PRD001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PRD Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRD001-101-J
Record Dates: First submitted 2025-03-27; First posted 2025-06-24 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1A: Single Ascending Dose (Experimental)
  Interventions: Drug: PRD001; Drug: Placebo
- Part 1B: Dietary effects (Experimental)
  Interventions: Drug: PRD001
- Part 2A: 14 days Multiple Ascending Dose (Experimental)
  Interventions: Drug: PRD001; Drug: Placebo
- Part 2B: 28 days Multiple Ascending Dose (Experimental)
  Interventions: Drug: PRD001; Drug: Placebo

INTERVENTIONS:
Drug: PRD001 — PRD001 capsules will be provided for oral administration
Drug: Placebo — Placebo capsules will be provided for oral administration
  Arms: Part 1A: Single Ascending Dose; Part 2A: 14 days Multiple Ascending Dose; Part 2B: 28 days Multiple Ascending Dose

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of PRD001 in healthy participants and to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of PRD001 in participants with borderline/mild hyper-LDL-cholesterolemia and mild fatty liver.

ELIGIBILITY:
Inclusion Criteria:

* Part 1A and Part 2A

  1. Healthy men aged between 18 and 45 years inclusive at the time of signing the informed consent form (ICF)
  2. Individuals who are willing and able to comply with the protocol schedule, including all scheduled visits, treatment plans, laboratory tests, and other trial procedures.
  3. Individuals who are able to participate in Part 1B following Part 1A, and are willing and able to comply with the protocol schedule, including all scheduled visits, treatment plans, laboratory tests, and other trial procedures.
  4. Individuals who have no clinically significant findings, are generally healthy and have no disease requiring medical treatment, based on medical history, physical examinations, vital signs, 12-lead ECG, and laboratory test results at screening.
  5. For Japanese participants in Part 1A and Part 2A, individuals whose parents and maternal and paternal grandparents are Japanese, and for Caucasian participants in Part 2A, individuals whose parents and maternal and paternal grandparents are Caucasian.
* Part 1B Individuals who receive PRD001 in Part 1A and complete all specified visit schedules.
* Part 2B

  1. Men aged between 18 and 60 years inclusive at the time of signing the ICF
  2. Individuals who are willing and able to comply with the protocol schedule, including all scheduled visits, treatment plans, laboratory tests, and other trial procedures.
  3. Individuals who have no clinically significant findings, are generally healthy and have no disease requiring medical treatment (however, diet or exercise therapy is acceptable), based on medical history, physical examinations, vital signs, 12-lead ECG, and laboratory test results at screening.
  4. Individuals whose parents and maternal and paternal grandparents are Japanese.
  5. Individuals who meet the following criteria:

     i. Individuals with mild-hyper-LDL-cholesterolemia ii. Individuals with mild hepatic steatosis

     Exclusion Criteria:
* All parts

  1. Individuals with active, latent, or inadequately treated M. tuberculosis infection at screening who meet both of the following:

     i. A positive result on the QuantiFERON-TB Gold test or an equivalent test ii. Active tuberculosis infection that is untreated, inadequately treated, or currently being treated
  2. Individuals with a history of human immunodeficiency virus (HIV) infection, syphilitic infection, hepatitis B or C at screening.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs and SAEs as assessed by vital signs | 42 days (treatment period: 28 days, observation period: 14 days)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Fukuoka, Japan